CLINICAL TRIAL: NCT02842476
Title: Accuracy Validation of the Cadwell Pulse Oximetry System
Status: Completed | Type: Observational
Sponsor: Cadwell Industries, Inc. (Industry)
Collaborators: Clinimark, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: PR 2016-177
Record Dates: First submitted 2016-07-15; First posted 2016-07-25 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Anoxia
Keywords: pulse oximetry
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Arterial blood samples were drawn during simultaneous data collection from the test devices. The blood was immediately analyzed by Reference CO-Oximetry providing functional SaO2 for the basis of the SpO2 accuracy comparison.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Disposable Sensor: Adhesive based Pulse Oximeter Probes, Model S0136J
  Interventions: Device: Disposable Sensor
- Reusable Sensor: Reusable Pulse Oximeter Probes, Model S0080D
  Interventions: Device: Reusable Sensor
- Control Pulse Oximetry: Reference CO-Oximeters ABL80 Flex OSM (Radiometer), # 302125, 307205 IL682 (Instrumentation Laboratories), # 012511B (ILH), #012511A (ILG)
  Interventions: Device: Control Pulse Oximetry

INTERVENTIONS:
Device: Disposable Sensor — Two adhesive based Pulse Oximeter Probes, S0136J-L were connected to the Cadwell Pulse Oximetry and then placed on each subject to evaluate the SpO2 accuracy performance during steady state non-motion conditions.
  Other Names: Model S0136J-L
  Groups: Disposable Sensor
Device: Reusable Sensor — Two soft reusable Pulse Oximeter Probes, Model S0080D-S were connected to the Cadwell Pulse Oximetry and then placed on each subject to evaluate the SpO2 accuracy performance during steady state non-motion conditions.
  Other Names: Model S0080D-S
  Groups: Reusable Sensor
Device: Control Pulse Oximetry — A Clinimark Control Pulse Oximetry system was also placed on the subject to evaluate the stability of the draws.
  Other Names: Reference Co-Oximeters, ABL80 Flex OSM (Radiometer): # 302125, 307205 IL682 (Instrumentation Laboratories): # 012511B (ILH), #012511A (ILG)
  Groups: Control Pulse Oximetry

SUMMARY:
The purpose of this study is to evaluate the SpO2 accuracy and performance of the Cadwell Pulse Oximetry system during non-motion conditions over the range of 70-100% SaO2 as compared to arterial blood samples assessed by CO-Oximetry for SpO2 validation. The end goal is to show the SpO2 accuracy performance of the Cadwell Pulse Oximetry System. It is expected that the Accuracy Root Mean Square (Arms) performance of the Cadwell Pulse Oximetry System will meet a specification of 3 or better in non-motion conditions for the range of 70-100% SaO2 thereby demonstrating an acceptable SpO2 accuracy performance specification.

DETAILED DESCRIPTION:
The SpO2 accuracy performance of the Cadwell Pulse Oximetry systems will be evaluated during non-motion conditions over the range of 70-100% SaO2 and compared to arterial blood samples assessed by COOximetry. A minimum of 10 healthy adult subjects, ranging in pigmentation from light to dark, will be enrolled in the study to meet the study design requirements defined by ISO 80601-2-61 and by the FDA's Guidance for Pulse Oximeters (March 4, 2013). The subjects will have an arterial catheter placed in the radial artery to allow for simultaneous blood samples during stable plateaus of induced hypoxic levels. The investigational devices will be placed on fingers for the test sites. Simultaneous data collection will be set up for each of the systems under test.

For the data analysis, the control oximeter will be used to assess the stability of each data point. Data that is found to be unstable will be removed prior to the comparative analysis. Next the CO-Oximeter data will be reviewed to make sure it does not contain any anomalous values such as elevated COHb, MetHb or inconsistent data. Anomalous values will be removed from the analysis prior to pairing of the SpO2 and SaO2 data. The statistical analysis is performed on a minimum of 200 data points collected on at least 10 subjects for the range of 67% to 100% SaO2. Functional SaO2 as measured by Reference CO-Oximetry will be used as the basis for comparison. The Accuracy Root Mean Square (ARMS) calculation is used to determine the SpO2 accuracy performance. Success will be achieved with an ARMS of 3 or better showing equivalence to the Gold Standard Reference CO-Oximetry providing documentation to support SpO2 accuracy claims for the investigational device.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and provide written informed consent
* 18 to 50 years of age
* Non-smoker or who has not smoked within 2 days prior to the study.
* Male or female
* Any race

Exclusion Criteria:

* Morbidly obese (defined as BMI >39.5)
* Compromised circulation, injury, or physical malformation of fingers, toes, hands, ears or forehead/skull
* Females who are pregnant, who are trying to get pregnant, or have a urine test positive for pregnancy on the day of the study
* COHb levels >3% as assessed with a Masimo Radical 7 (Rainbow)
* Respiratory conditions
* Heart or cardiovascular conditions
* Self reported health conditions
* Blood clotting disorders
* Severe contact allergies to standard adhesives, latex or other materials
* Unwillingness or inability to remove colored nail polish from test digits
* Other known health condition, should be considered upon disclosure in health

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Following Salus Independent Review Board (IRB) approval for the Study Procedure Title: "Accuracy Validation of the Cadwell Pulse Oximetry System", Clinimark Study ID# PR 2016-177, eleven healthy adult volunteer subjects were enrolled into the study. The demographics for the study included five males and six females (age: 21-46yrs, weight: 118-220lbs, height: 60-74", BMI: 20.9-30.7). For the demographics based on race, the subject pool included one Black / African-American, three Asians (one of Indian descent), and seven White. The ethnicity for the group is four Hispanic, and seven Non-Hispanic / Non-Latino. The skin pigmentation / tones ranged from light to dark meeting the requirement of at least 2 darkly pigmented or 15 % of the subject pool whichever is larger.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2016-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
SpO2 Sensor Values | Through study completion, an average of 1 day
  SpO2 values (%) from the Cadwell pulse oximetry device using disposable and reusable sensors were collected electronically at one second intervals.

SECONDARY OUTCOMES:
Arterial Oxygen Saturation | Through study completion, an average of 1 day
  Each subject was presented with various levels of induced hypoxia resulting in stable oxygen saturation levels between 100% and 67% SaO2. Arterial blood draws were collected under non-motion conditions. The blood was immediately analyzed to measure the arterial oxygen saturation.

IPD SHARING:
Plan to Share IPD: No